CLINICAL TRIAL: NCT01154738
Title: Influence of Lidocaine on a Closed-Loop Anesthesia System
Brief Title: Lidocaine and Closed-Loop Anesthesia System
Acronym: LoopLido
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/18; 2010-019979-29 (EudraCT Number)
Record Dates: First submitted 2010-06-25; First posted 2010-07-01 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and Lidocaine
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): patients will receive a closed-loop administration of propofol and remifentanil according to bispectral level and a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — bolus dose of lidocaine (1.5 mg.kg-1) followed by an infusion of lidocaine (2 mg.kg-1 h-1) until the end of anesthesia.
  start of the induction of anesthesia 10 minutes after the bolus dose of lidocaine
  Arms: Lidocaine
Drug: Placebo — NaCl 9/00 (same volume as in the lidocaine group)
  start of the induction of anesthesia 10 minutes after the bolus dose of NaCl 9/00
  Arms: Placebo

SUMMARY:
The objective is to evaluate the sparing effect of Lidocaine on doses of propofol and remifentanil.

ELIGIBILITY:
Inclusion Criteria:

* patients ASA 1, 2 or 3 scheduled for a general anesthesia surgical procedure (abdominal surgery, urology, ENT major procedure) lasting between 1 and 3 hours

Exclusion Criteria:

* age under 18 years
* simultaneous general and loco-regional anesthesia
* allergy to NSAID
* treatment with verapamil, ketamine or gabapentin
* patients receiving an opioid preoperatively
* severe hepatic insufficiency
* contra-indication to lidocaine
* contra-indication to propofol or to remifentanil
* history of central nervous system disease
* patients receiving a psychotropic treatment
* patients with a pace-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
administered dose of propofol during maintenance of anesthesia | day 1

SECONDARY OUTCOMES:
administered dose of propofol during induction of anesthesia | day 1
administered doses of remifentanil during induction and maintenance of anesthesia | day 1
delay (measured as minutes) between the end of propofol and remifentanil administration and the recovery from anesthesia | day 1
hemodynamic abnormalities requiring treatment | day 1
% of time with a BIS index between 40 and 60 | day 1
postoperative morphine requirement | day 1
incidence of postoperative nausea and vomiting | day 1
% of patients with an explicit memorisation of the intraoperative period | second postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, Study Chair — Hôpital Foch
Locations (1):
- Hopital Tenon, Paris, France